CLINICAL TRIAL: NCT03418610
Title: Azelaic Acid Foam 15% in the Treatment of Papulopustula Rosacea: An Evaluation of Photographic Evidence
Brief Title: Azelaic Acid Foam 15% in the Treatment of Papulopustular Rosacea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Research Center of the Carolinas (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bayer Rosacea
Record Dates: First submitted 2017-12-12; First posted 2018-02-01 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2018-01

CONDITIONS: Rosacea, Papulopustular
Keywords: Rosacea
MeSH Terms: conditions — Rosacea | interventions — azelaic acid

STUDY DESIGN:
Intervention Model Description: Single Site, Single Arm Open Label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open Label Single Arm (Other): Azelaic Acid Foam 15% applied twice daily
  Interventions: Drug: Azelaic Acid foam 15%

INTERVENTIONS:
Drug: Azelaic Acid foam 15% — mild to moderate rosacea
  Other Names: Finacea

SUMMARY:
This research study is being performed to evaluate the photographic evidence of the efficacy and tolerability of Azelaic Acid Foam 15% in the treatment of papulopustular rosacea.

DETAILED DESCRIPTION:
This is a single site, single arm open label study of Azelaic Acid foam 15% for the treatment of moderate to severe papulopustular rosacea. All patients will apply Azelaic Acid foam twice daily. At scheduled visits, high resolution equipment will be used to measure 3D topographical values for elevation of papules and pustules to objectively evaluate reduction of papulopustular lesions. Investigator and subject assessments will also be completed to assess the level of rosacea at weeks 4,8 and 12.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age 18 or older.
2. Diagnosis of moderate to severe papulopustular rosacea with IGA of 3- moderate or 4-severe.
3. Presence of 12 - 50 inflammatory lesions and persistent erythema with or without telangiectasia.
4. Subjects must read, understand, and sign the Informed Consent.
5. Subjects must be willing and able to comply with study procedures and visit schedule requirements.
6. Women of childbearing potential that are willing to use an acceptable method of contraception during the study.

Exclusion Criteria:

1. Active or localized or systemic infections.
2. Subjects must not be immunocompromised.
3. Known unresponsiveness or allergy to azelaic acid.
4. Subjects unlikely to comply with the protocol, e.g. mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the clinical study, uncooperative attitude or unlikelihood of completing the study (e.g. drug or alcohol abuse).
5. Subjects must not be pregnant or breastfeeding.
6. Presence of dermatoses that might interfere with the ability to diagnose and/or evaluate rosacea.
7. Presence of other types of rosacea.
8. Laser surgery on the face for the treatment of telangiectasia or other conditions within 6 weeks of study enrollment.
9. Use of medications or products for the treatment of rosacea or other medical conditions within the following time periods prior to study enrollment. Use of these medications will be prohibited during the trial.

   Topical Prescription or Nonprescription medications 6 weeks Oral retinoids 6 months Tetracycline (ex. doxycycline, minocycline 2 months Corticosteroids 4 weeks Erythromycin or azithromycin 4 weeks Other systemic medications to treat rosacea 6 weeks
10. Refusal to sign the Informed Consent document or Photo Release document and/or refusal to comply with all follow-up requirements.
11. Use of medications that are known to cause flushing.
12. Dose changes in the last 90 days or initiation of beta-blockers, vasodilators, vasoconstrictors, nonsteroidal anti-inflammatory drugs, hormone therapy, and/or other drugs known to cause acneform eruptions.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
Inflammatory Lesion Count | 12 weeks
  The change in inflammatory lesion counts at week 12 compared to baseline

SECONDARY OUTCOMES:
Investigator Global Assessment | 12 weeks
  Severity of Disease by Investigator Global Assessment, Score of 0 (Clear) - 4(Severe)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Schlesinger, MD, FAAD, Principal Investigator — Medical Director
Locations (1):
- Clinical Research Center of the Carolinas, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided